CLINICAL TRIAL: NCT02231424
Title: Postmarketing Surveillance Study (as Per § 67 (6) AMG [German Drug Law]) of Berodual® Metered-dose Inhaler in Chronic Obstructive Airways Disease
Brief Title: Postmarketing Surveillance Study of Berodual® Metered-dose Inhaler in Chronic Obstructive Airways Disease
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 215.1353
Record Dates: First submitted 2014-09-01; First posted 2014-09-04 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — fenoterol, ipratropium drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- chronic obstructive respiratory tract disease patients
  Interventions: Drug: Drug: Berodual®

INTERVENTIONS:
Drug: Drug: Berodual®

SUMMARY:
The aim of this postmarketing surveillance is to obtain further information about the tolerability and efficacy of Berodual® metered-dose inhaler in the treatment of chronic obstructive respiratory tract disease under conditions of daily practice

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex, including children over 6 years
* Chronic obstructive respiratory tract disease. Every doctor was asked to include in this study the first patients coming after each other, who were treated for the first time with Berodual® metered dose inhaler (MDI)

Exclusion Criteria:

* Contraindications listed in the Instructions for Use/Summary of Product Characteristics of Berodual® metered-dose inhaler

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diagnosis of chronic obstructive respiratory tract disease
Sampling Method: Non-Probability Sample
Enrollment: 713 (Actual)
Dates: Start 1999-01; Primary Completion 1999-11 (Actual)

PRIMARY OUTCOMES:
Overall severity of the clinical picture rated on a 4-point scale | after 3 and 6 weeks

SECONDARY OUTCOMES:
Changes in dyspnea and/or asthma attacks rated on a 4-point scale | after 3 and 6 weeks
Number of dyspnea episodes rated on a 4-point scale | after 3 and 6 weeks
Number of awakenings due to night-time dyspnea rated on a 4-point scale | after 3 and 6 weeks
Assessment of morning coughing with expectoration rated on a 4-point scale | after 3 and 6 weeks
Assessment of tolerability on a 4-point scale | after 3 and 6 weeks
Number of patients with adverse drug reactions | up to 6 weeks
Changes in pathological auscultation findings rated on a 3-point scale | after 3 and 6 weeks
Changes in concomitant medication | up to 6 weeks
Assessment of efficacy on a 4-point scale | after 3 and 6 weeks